A Phase II Double-blind, Randomised, Parallel Group 2:1
Comparison of the Efficacy and Safety of FP-1201-lyo
(Recombinant Human Interferon beta-1a) and Placebo in
the Prevention of Multi-Organ Failure on Patients Surviving
Open Surgery for a Ruptured Abdominal Aortic Aneurysm

NCT03119701

SAP Version: Final

SAP Date: 19 Dec 2019

A Phase II Double-blind, Randomised, Parallel Group 2:1 Comparison of the Efficacy and Safety of FP-1201-lyo (Recombinant Human Interferon beta-1a) and Placebo in the Prevention of Multi-Organ Failure on Patients Surviving Open Surgery for a Ruptured Abdominal Aortic Aneurysm

Study code: INFORAAA

Phase II study

STATISTICAL ANALYSIS PLAN

# **Signatures:**

Statistical Analysis Plan was prepared by:



Statistical Analysis Plan was reviewed/approved by:



## **Table of Contents**

| 1 | Abbreviations | 4 |
|---|---|---|
| 2 | General remark | 4 |
| 3 | Study objective(s) | 4 |
| 4 | Design and type of the study | 5 |
| 5 | Study variables | |
| 6 | Sample size considerations | |
| 7 | Statistical hypotheses | |
| 8 | Analysis datasets | |
| 9 | General statistical considerations. | |
| 9. | | |
| 9. | .2 Handling of drop-outs or missing data | |
| 9. | .3 Interim analyses and data monitoring | 8 |
| | .4 Multicenter studies | |
| | .5 Multiple comparison/multiplicity | |
| | .6 Examination of subgroups | |
| 10 | Demographic and other baseline characteristics | |
| 11 | Extent of exposure and compliance | |
| 12 | Analysis of efficacy | |
| | 2.1.1 Primary efficacy variables | |
| | <ul><li>2.2 Secondary efficacy variables</li><li>2.3 Additional analyses</li></ul> | |
| | <ul><li>2.3 Additional analyses</li><li>2.3.1 Pharmacodynamics and tentative disease specific marker analysis</li></ul> | |
| | 2.3.2 Pharmacoeconomic analysis | |
| 13 | Ţ | |
| | 3.1 Adverse events | |
| 13 | 3.2 Laboratory safety variables | |
| 13 | 3.3 Other safety variables | 13 |
| 14 | Completion and premature discontinuation | 13 |
| 15 | Deviations from the analyses planned in the study protocol | 13 |
| 16 | Execution of statistical analyses | 14 |
| 17 | Hardware and software | |
| 18 | References | |
| 19 | Appendices | |
| | 9.1 Study flow chart | |
| | 9.2 Study procedure flow charts | |
| | 9.3 Table and figure plan | |
| 19 | 9.4 Data listing plan | 24 |

#### 1 Abbreviations

AE Adverse event

ANOVA Analysis of variance

ATC Anatomical Therapeutic Chemical

FAS-E Full analysis set for efficacy
FAS-S Full analysis set for safety
IAP Intra-abdominal pressure

ICU Intensive care unit

MedDRA Medical dictionary of regulatory authorities

mRS Modified ranking scale
NAb Neutralizing antibody
PD Pharmacodynamics

PIM Potential Inflammatory Markers

PPS Per protocol set

SD Standard deviation
SAE Serious adverse event

SOFA Sequential organ failure assessment
TEAE Treatment emergent adverse event

VFD Ventilator free day

#### 2 General remark

This SAP version further details the SAP dated 17.6.2019, which was generated before performing the Interim analysis for the 35 evaluable patients. Study was discontinued after the Interim analysis. The earlier version of the SAP concentrated on the primary analyses and this version will entail all planned analyses. The analysis plans concerning the primary analyses are not changed from the previous version.

As the study was discontinued, analyses described here, will be performed on the available data gathered thus far.

## 3 Study objective(s)

The primary objective of this study is to evaluate the safety and the efficacy of FP-1201-lyo over placebo on all-cause mortality at study day 30; D30 (30 days from the first dose of study medication).

The secondary objectives of this study are

- 1. To evaluate the efficacy of FP-1201-lyo treatment by assessing short term outcomes (D30) and mid-term outcomes (D90 [3 months])
- 2. To evaluate the safety and tolerability of FP-1201-lyo treatment

- 3. To evaluate the pharmacodynamics (PD) of FP-1201-lyo
- 4. To evaluate the Tentative Disease Specific Marker CD73 and Potential Inflammatory Markers (PIM) IL-6 and HGF
- 5. To evaluate neutralizing antibodies against IFN beta-1a (NAbs)

### 4 Design and type of the study

This is a multicentre, randomised, double-blind, Phase II, parallel group comparison study of the efficacy and safety of FP-1201-lyo compared to placebo in patients surviving emergency open surgery for an infra-renal ruptured abdominal aortic aneurysm. Both treatment groups will receive standard supportive care.

Patients will receive  $10 \mu g$  FP-1201-lyo or placebo intravenously as a bolus injection once every 24 hours. The maximum duration of treatment will be 6 days. Treatment may be discontinued before 6 days if the patient's condition improves beyond the need for ICU treatment and if, in the opinion of the Investigator, the patient would likely not benefit from continuation of treatment.

With an estimated screening failure rate of approximately 15%, a maximum of 180 patients were planned to be consented and entered into the study in order to randomise and initiate treatment of 152 patients.

Study was discontinued after an Interim analysis.

### 5 Study variables

The following variables will be evaluated

### The demographic and baseline variables

Gender, age at entry, race, weight (predicted or actual), height, medical history, concomitant medications/therapies, major surgical outcomes affecting patient and pregnancy test (females of child bearing potential, and peri procedural information (duration of the surgical procedure for RAAA, total clamping time, total bleeding volume, total volume substitution, total blood substitution, total red blood cells substitution, total platelets substitution, total crystalloids substitution and total diuresis volume during procedure and recycling of blood during surgery (yes/no)).

### The primary efficacy outcome variable

- All-cause mortality at D30

### The secondary efficacy outcome variables

- All-cause mortality at D90 (3 months)
- Number of ventilator free days (VFDs) at D30
- Number of days receiving haemodialysis at D30 and D90
- Number of organ failure free days up to D30 by means of the SOFA score
- Prevalence of abdominal compartment syndrome, i.e. intra-abdominal pressure (IAP) between treatment groups
- Neutralizing antibodies against IFN beta (NAbs) in whole blood samples up to D30

- Disability on D90 measured by modified ranking scale (mRS)

### Safety variables

Adverse events, vital signs (body temperature, blood pressure, heart rate), physical examination and clinical laboratory parameters (biochemistry and haematology).

### Pharmacodynamic (PD) and tentative disease specific marker variables

- MxA (protein) concentration in whole blood samples from baseline up to D13
- CD73 concentration in serum samples from baseline up to D6
- Potential Inflammatory Markers (IL-6 and HGF) in serum samples from baseline up to D13

#### Pharmacoeconomic variables

- Length of ICU stay, in terms of ICU free days at D30
- Length of hospital stay, in terms of hospital free days at D90
- Length of stay at another health care facility at D90
- Length of haemodialysis needed

### 6 Sample size considerations

The primary efficacy endpoint is all cause mortality at D30. Death within 36 hours from the first dose of the study treatment leads to exclusion from efficacy analysis. A sample size of 129 eligible patients for the primary efficacy analysis, with a 2:1 ratio to active (86) and placebo (43), will detect the difference of 22% between the two treatment groups with 80 % power using 2-sided z-test with 0.05 significance level. To take account of the planned interim analysis, calculations assume that 2 sequential tests are made (in addition to final analysis) and the O'Brien-Fleming spending function is used to determine the test boundaries. Statistical analysis plan for the interim analyses will be presented in a separate document.

Power calculation assumes 37 % proportion of events on placebo group and 15 % proportion for the active treatment group.

To achieve a sample size of 129 for the primary efficacy analysis, taking account the estimated amount of early deaths within 36 hours from first dose of the study treatment (estimated 15 %), there should be 152 patients randomised to the study.

Study was discontinued after the first Interim analysis. Therefore, the sample size did not reach the 129 patients aimed for.

### 7 Statistical hypotheses

The primary objective of this study is to evaluate the safety and the efficacy of FP-1201-lyo over placebo on reducing all-cause mortality at study day 30, i.e., the null-hypothesis to be tested is

H<sub>0</sub>: FP-1201-lyo is not superior to control with respect to all-cause mortality at study day 30

against

H<sub>1</sub>: FP-1201-lyo is superior to control with respect to all-cause mortality at study day 30

#### 8 Analysis datasets

Statistical analyses will be performed on the following analysis datasets.

The Full Analysis Set for Efficacy (FAS-E) consists of all randomised patients receiving study treatment but excluding the early deaths (within 36 hours from first dose of study treatment) and comprises the analysis set on which the primary efficacy analysis is based.

The Per Protocol Set (PPS) consists of the patients in the FAS-E excluding patients with major protocol violations possibly affecting the primary study endpoint analysis.

The precise definition of the PPS at the patient level was planned to be identified at the blind review conducted both before the second interim and final analysis. The detailed criteria for patient classification will be prepared before database lock. Subject classification was to be created first for the subjects included in the second interim analysis, and later amended for the final analysis with the subjects that were not included in the interim analysis.

The first Interim analysis (after 35 evaluable patients) was based on FAS-E dataset. No classification for PPS was done for the first Interim analysis.

Statistical analyses for efficacy, PD, tentative disease specific markers and pharmacoeconomic variables are performed on both the FAS-E and PPS.

Study was discontinued after the first interim analysis. Subject classification document defining the analysis datasets in detail will be prepared and signed before database lock.

The Full Analysis Set for Safety (FAS-S) consists of all randomised patients receiving study treatment and comprises the analysis set on which the evaluation of safety is based. All safety analyses are performed on the FAS-S analysis dataset.

#### 9 General statistical considerations

Summary statistics will include at least the number of subjects, mean, standard deviation, median, minimum and maximum for continuous variables, and frequencies and percentages for categorical variables. All data collected will be listed by subject.

In the statistical analyses a p-value less than 0.05 will be considered as an indication of statistical significance. If not stated otherwise, all tests will be performed as two-sided tests and two-sided 95% confidence intervals will be produced. Missing values will not be imputed in the analyses.

#### 9.1 Adjustment for covariates

The primary model will include the stratification factors (age group and gender) used in the randomisation as covariates.

### 9.2 Handling of drop-outs or missing data

Missing values will not be imputed. Primary endpoint is mortality at Day 30 and all evaluable patients will be included in the primary analysis.

### 9.3 Interim analyses and data monitoring

Two Interim analyses were planned for the study with futility and efficacy stopping criteria using O'Brien-Fleming boundaries.

Study was discontinued after the first interim analysis.

#### 9.4 Multicenter studies

Handling of centers was to be defined before second interim analysis when there would be better understanding of the center size.

Study was discontinued after the first interim analysis. Patient accrual to the different study centers was varying in amounts. Center info will not be used directly in the analyses, but country and site will be included in the tabulations of patient demographics.

### 9.5 Multiple comparison/multiplicity

There is one primary efficacy variable in the primary hypothesis of this study; all-cause mortality at D30. The primary evaluation of this hypothesis will be based upon the FAS-E dataset. This in itself will not give reason to adjustments for multiple comparison/multiplicity.

However, two interim analyses were to be performed after reaching 35 and 84 evaluable patients for the primary efficacy variable. For this reason, the primary efficacy endpoint was to be evaluated using O'Brien and Fleming criteria controlling the type I error rate. Using the O'Brien-Fleming spending function on the two sequential tests will cause the nominal alpha level for the primary efficacy variable in final analysis to be 0.04664. Therefore, for the primary efficacy variable a p-value less than 0.04664 will be considered as statistically significant.

As the study was discontinued after the first interim analysis, the planned O'Brien and Fleming correction will not be applied to the primary analysis. Instead, the standard p-value of less than 0.05 will be considered statistically significant.

#### 9.6 Examination of subgroups

Data for the primary efficacy endpoint will also be presented for key, pre-defined subgroups of patients. Concomitant use of glucocorticoids will be one key subgroup as earlier studies have suggested that it may have effect on the study treatment. As CD73 response (and IL-6 and HIF-1 $\alpha$ ) may be also genetically determined/individual, another key subgroups will be CD73 responder status (determined by a 2-fold elevation in CD 73 (from baseline to peak value). In addition, if analyses indicate yet another, but currently unknown but relevant subgroups, they will be analysed as separate subgroup analyses for exploratory purposes

Key subgroups included in analyses

- Concomitant use of glucocorticoids
- CD 73 responder status (responders vs. non-responders)
- IL-6 responder status
- HIF- $1\alpha$  responder status

### 10 Demographic and other baseline characteristics

Number of patients enrolled into the study at screening and the reasons for screening failures will be summarized. The number of patients entering and completing the study will be summarized. All patients discontinuing the study will be summarized together with the reason(s) for discontinuation.

Demographic and baseline characteristics will be summarized by treatment using descriptive statistics. Following variables will be analysed.

- Gender
- Age at entry
- Race
- Height
- Weight
  - o If actual weight is not available for a patient, then predicted body weight will be used in its place
  - o Predicted body weight (kg) is calculated using the following formulae:
    - Males: 50 + 0.91 (height in cm 152.4)
    - Females: 45.5 + 0.91(height in cm 152.4)
- Major surgical outcomes affecting patient
  - Open abdomen (yes/no)
  - o Left renal vein ligated (yes/no)
  - o Clamping time above the renal arteries
- Medical history
- Concomitant medications/therapies
- Pregnancy test (females of child bearing potential).

Similarly, the duration of the surgical procedure and peri procedural information will be summarized by treatment. Additional concomitant procedures will be listed only.

Medical history and concomitant medications/therapies will be presented only by frequency and subject count-based tables according to WHO Anatomical Therapeutic Chemical (ATC) classification.

Pregnancy test results (females of child-bearing potential) will be presented only descriptively by a subject count-based table.

### 11 Extent of exposure and compliance

Treatment exposure, study duration and treatment compliance will be summarised by treatment groups using descriptive statistics.

### 12 Analysis of efficacy

### 12.1.1 Primary efficacy variables

Primary efficacy variable is the all-cause mortality at D30. The primary efficacy analysis will be conducted using logistic regression model for the observed mortality rates in the two treatment groups. Stratification factors sex and age used in the randomisation will be included in the model. Primary result will be presented as an adjusted odds ratio and a 95% CI for the adjusted odds ratio. Also, a 95% exact unconditional confidence interval (CI) for the difference in the observed mortality rates will be calculated. As a sensitivity analysis, unadjusted results will also be presented.

For the primary comparison, a p-value less than 0.04664 was planned to be considered as statistically significant due to O'Brien-Fleming alpha spending used for the Interim analyses. Due to the study discontinuation after the first Interim analysis, two-sided significance level of 0.05 will be used for all analyses.

### 12.2 Secondary efficacy variables

The following secondary endpoints will be analysed:

- Time and reason/diagnosis of death up to D90 (3 months)
- Number of VFDs up to D30
- Number of days receiving hemodialysis at D30\*
- Number of ICU free days up to D30\*
- Organ failure free days up to D30
- Number of days in hospital up to D30 (length of stay in another

health care facility)\*

• Prevalence of abdominal compartment syndrome, i.e. intra-abdominal pressure

(IAP) value differences between study groups

- Disability on D90 measured by modified ranking scale (mRS)
- Neutralizing (and anti-drug) antibodies IFN beta (ADAs and NAbs) in whole blood samples up to D30

\*ICU free days and number of days in hospital, length of stay in another health care facility and number of days receiving hemodialysis at D90 summarized in pharmacoeconomic tables

All-cause mortality at D90 (3 months) will be compared using Cox regression model including stratification factors (if feasible). Estimated hazard ratios will be presented with associated 95% CIs and log-rank p-values for the FAS-E. Also, similar logistic regression as for the primary endpoint (D30 mortality) will be done.

For endpoints number of VFDs, number of ICU free days, organ failure-free days, number of days on hemodialysis, number of days in hospital, length of stay in another health care facility and IAP values, data will be summarised in terms of the mean, median, minimum and maximum, and the treatment groups will be compared using the Mann-Whitney U-test. Descriptive tables of IAP grade by timepoint will be presented using counts and percentages. Number of days on hemodialysis, number of days in hospital, length of stay in another health care facility and IAP value analyses will be performed for all patients and excluding deaths separately.

Complete data on organ failure free days may be unavailable due to SOFA scores not being assessed after ICU treatment. To account for this, the number of organ failure free days will be analysed by expressing these as a proportion of the days on which SOFA scores are available.

Disability measured with mRS will be summarized descriptively and the treatment groups will be compared using the Cochran-Mantel-Haenszel test for trend.

ADAs and NAbs in whole blood samples up to D30 will be summarized using descriptive statistics.

All secondary analyses are designed to be supportive of the analysis of the primary endpoint and there will be no adjustments for the multiplicity of endpoints so that each analysis will be undertaken at the two-sided 5% level of significance.

### 12.3 Additional analyses

Additional analyses are performed on PD and tentative disease specific marker variables and pharmacoeconomic variables.

#### 12.3.1 Pharmacodynamics and tentative disease specific marker analysis

PD and tentative disease specific marker variables to be analysed are MxA concentration in whole blood samples from baseline up to D13, CD73 concentration in serum samples from baseline up to D6 and potential Inflammatory Markers (e.g. IL-6 and HIF-1α) in serum samples from baseline up to D13.

These will be summarised using descriptive statistics and analysed using Repeated measurements ANOVA model with main effects of treatment and day and their interaction. Correlations between the repeated observations will be modelled using compound symmetry covariance structure. The model will be used to estimate population geometric means (95 % CI) for the treatment groups by timepoint.

### 12.3.2 Pharmacoeconomic analysis

Following pharmacoeconomic endpoints were defined for the study:

- Length of ICU stay, in terms of ICU free days at D90
- Length of hospital stay, in terms of hospital free days at D90
- Length of stay at another health care facility at D90
- Length of hemodialysis needed (at D90)

Due to early discontinuation of the study, these endpoints will not be analysed.

### 13 Analysis of safety and tolerability

All subjects in the SAF-S analysis set (all randomised patients receiving study treatment) will be included in the safety and tolerability analysis. Safety variables to be analysed are; adverse events, clinical laboratory parameters, vital signs and physical examination.

#### 13.1 Adverse events

All recorded adverse events will be coded according to the Medical Dictionary for Regulatory Activities (MedDRA). Treatment emergent adverse event (TEAE) is defined as an AE that begins or worsens in severity after at least one dose of study drug has been administered. Non-treatment emergent AEs are listed only.

TEAEs will be summarized using frequency and subject based tables. TEAEs will be tabulated by treatment group, system organ class (SOC), preferred term (PT), causality and severity. For analysis purposes, each subject will also be categorized by the maximum severity reported for a given TEAE and these will be tabulated by maximum severity. TEAEs will be summarized separately for treatment period (D1-D5) and short-term follow-up period (D6-D30). TEAEs are not collected, and therefore not reported, during the mid-term follow-up.

Serious adverse events (SAEs) and AEs leading to discontinuation will be summarized by treatment groups. All deaths up to D90 are reported as SAEs.

### 13.2 Laboratory safety variables

Laboratory safety variables (biochemistry and haematology) to be analyzed are presented in table 1 below. Descriptive statistics and the frequency and percentage of absolute values below, within and above the reference range will be tabulated for the safety laboratory variables at D0 (baseline), D1, D2, D3, D4, D5, D6, D9, D13 and D30. Descriptive statistics will include mean, median, standard deviation (SD), minimum and maximum.

In addition, shift tables (within, below and above the normal range) will be provided for each parameter in relation to the maximum change from baseline from D0 over the complete 30-day follow-up period.

Table 1. Laboratory Variables

| Biochemistry | Haematology Includes coagulation |
|---|---|
| Alanine transaminase (ALAT) Alkaline phosphatase (AFOS) Aspartate transaminase (ASAT) Bicarbonate Lactate pH Bilirubin Calcium Creatinine Potassium Sodium (blood gas value acceptable) | Hemoglobin Leucocyte differential count (absolute) Mean cell volume Platelet count Red cell count White cell count |

### 13.3 Other safety variables

Other safety variable to be analysed are vital signs (body temperature, blood pressure, heart rate) and physical examination.

Vital signs data is summarized by treatment groups separately at D0, D1, D2, D3, D4, D5, D6, D9, D13 and D30. Absolute values and changes from baseline are both summarized. In addition, the maximum change from baseline over the 30-day follow-up period will be calculated for each patient and summarized. Vital signs summaries will be in terms of mean, median, SD, minimum and maximum.

Physical examination covering all the major organ systems will be performed at screening and D30. These will be summarized by treatment groups and visits using frequency and percentage of normal/abnormal observations. In addition, shift tables will be provided describing the change from screening to D30.

### 14 Completion and premature discontinuation

Completion and premature discontinuation will be listed. The reasons for premature discontinuation will be presented.

### 15 Deviations from the analyses planned in the study protocol

Study was discontinued after the first Interim analysis. Due to the early discontinuation, the planned O'Brien and Fleming correction will not be applied to the primary analysis. Instead, the standard p-value of less than 0.05 will be considered statistically significant.

Due to low number of accrued patients, the center effect was not further explored in the analyses. Analysis of study centers was limited to summary statistics for baseline information.

Due to the early discontinuation of the study, the pharmacoeconomic endpoints (see section 12.3.2) will not be analysed.

There are no other major deviations in the statistical analysis plan from the analyses planned in the study protocol.

### 16 Execution of statistical analyses

Statistical analyses will be performed by

### 17 Hardware and software

Statistical analysis, tables and patient data listings will be performed with SAS® version 9.4 or later for Windows (SAS Institute Inc., Cary, NC, USA).

#### 18 References

Clinical Study Protocol (FP1CLO006), Final Protocol version 05 (16 April 2019), Faron Pharmaceuticals Ltd.

### 19 Appendices

### 19.1 Study flow chart



# 19.2 Study procedure flow charts

# Flow chart for Baseline and Treatment periods

| | Baselin | e Period | 58 | | Treatmen | nt Period* | | |
|---|---|---|---|---|---|---|---|---|
| ASSESSMENTS | Screen | D0 | D0 | D1 | D2 | D3 | D4 | D5 |
| | Enrolment | pre-dose | ICU | | | | | |
| Symptoms, diagnosis and treatment of RAAA | X | | | | | | | |
| Medical History | X | 3 | | | | | | |
| Inclusion / Exclusion Criteria | X | | | | | | | |
| Confirmation of all eligibility criteria | | X | | | | | | |
| Informed Consent + | X | | | | | | | |
| Demography | X | , | | | | | | |
| Physical Exam (incl. PB, pulse) | X | | | | | | | |
| Time of onset of symptoms | Х | | × | | | | | |
| Hemodynamic collapse before ER | X | | | | | | | |
| Date and time of entry to ER | X | | | | | | | |
| Moving to OR for open repair | X | -3 | | | | | | |
| Patient Randomisation (after consent & elig bility criteria confirmed) | | х | | | | | | |
| Hemodynamic collapse before clamping (yes/no) | | х | | | | , | | |
| Proximal aortic clamp used(minutes/no) | | X | | | | | 20 | |
| Check that renal arteries are intact | | X | | | | | | |
| Check that RAAA is infrarenal | | X | | | | | | |
| Check that the patient is still salvageable, no irreversible shock | | х | X | | | | | |
| mRS | | X | | | | * | | |
| SOFA Scoring <b></b> (the worst obtained daily value should be used) | | | X | <b>X</b><br>6-10am | <b>X</b><br>6-10am | <b>X</b><br>6-10am | <b>X</b><br>6-10am | <b>X</b><br>6-10am |
| Ventilator Free Days (VFDs) | Í | | X | X | X | X | X | X |
| Vital Signs; Temp, BP, HR (closest to 8am) | | х | | <b>X</b><br>6-10am | <b>X</b><br>6-10am | <b>X</b><br>6-10am | <b>X</b><br>6-10am | <b>X</b><br>6-10am |
| Blood Biochemistry | | X | | <b>X</b><br>6-10am | <b>X</b><br>6-10am | <b>X</b><br>6-10am | <b>X</b><br>6-10am | <b>X</b><br>6-10am |
| Haematology | | X | | <b>X</b><br>6-10am | <b>X</b><br>6-10am | <b>X</b><br>6-10am | <b>X</b><br>6-10am | <b>X</b><br>6-10am |
| Intra-abdominal pressure (IAP) | | | | <b>X</b><br>6-10am | <b>X</b><br>6-10am | <b>X</b><br>6-10am | <b>X</b><br>6-10am | <b>X</b><br>6-10am |
| FP-1201-lyo or placebo<br>administration⊽ | | | Dose1 | Dose 2 | Dose 3 | Dose 4 | Dose 5 | Dose 6 |
| MxA, CD73 and PIM | | X<br>1h<br>pre-dose | | X<br>22h ±2h<br>since | X<br>22h ±2h<br>since | X<br>22h ±2h<br>since | X<br>22h ±2h<br>since | X<br>22h ±2h<br>since |
| | | | | Dose2 | Dose 3 | Dose 4 | Dose 5 | Dose 6 |

| Concomitant Medications/Therapies | X | X | X | х | X | X | х | X |
|---|---|---|---|---|---|---|---|---|
| AE Recording (after obtained consent) | | x | X | x | х | х | x | x |
| Major surgical outcome recording | | | X | X | X | X | X | X |
| Assessment of mortality and reason/diagnosis of death | х | x | x | x | х | х | х | x |

### KEY:

- \* Assessments prior to D30 are only performed if patient is still hospitalised in the same hospital initially operated. If the patient is moved to a different hospital, assessements will not be done. If study treatment is terminated early by Investigator decision due to patient improvement, the study assessment schedule should be followed as normal.
- + Study specific procedures must be performed after informed consent for the study is obtained. If ICU standard procedures are in line with the study procedures and if the timing of RAAA diagnosis, consent, operative treatment and dosing preclude repetition of procedures for the purposes of the study, then standard patient care test results may be used for screening even prior to obtaining consent
- ∇ Study medication, FP-1201-lyo or placebo is administered as a bolus intravenous injection, followed by a 5 ml flush of sterile saline. On D0 the first dose of study medication is administered at 0h. Subsequent doses from D1 to D5 are administered every 24 hours ± 1 hour.
- SOFA scores are assessed daily in the ICU from D1 to D30, as applicable by standard clinical treatment at that point (therefore if a patient doesn't have an arterial line, no arterial blood sampling should be taken)

#### Flow Chart for the Short Term and Mid Term Follow-up Periods

| | | Short Term Follow-Up* | | | |
|---|---|---|---|---|---|
| ASSESSMENTS | D6 | D9** | D13** | D30 | D90<br>(+14 days)<br>3 months |
| Check whether patient is in the ICU | х | X | x | x | |
| Check whether patient is on ventilation | x | x | x | x | |
| Check whether patient is on organ support (hemodialysis) | х | X | X | х | х |
| SOFA Scoring <b>*</b> (worst daily value should be used) | х | x | x | х | |
| Ventilator Free Days (VFDs) | х | x | х | х | |
| Physical Examination | х | X | х | x | o 8 |
| Vital Signs; Temp, BP, HR<br>(closest to 8am) | <b>X</b><br>6-10am | <b>X</b><br>6-10am | <b>X</b><br>6-10am | <b>X</b><br>6-10am | |
| Blood Biochemistry | <b>X</b><br>6-10am | <b>X</b><br>6-10am | <b>X</b><br>6-10am | <b>X</b><br>6-10am | |
| Haematology | <b>X</b><br>6-10am | <b>X</b><br>6-10am | <b>X</b><br>6-10am | <b>X</b><br>6-10am | |
| Intra-abdominal pressure (IAP) | <b>X</b><br>6-10am | <b>X</b><br>6-10am | <b>X</b><br>6-10am | | |
| MxA, CD73 and PIM | X<br>22h±2h<br>since Dose 6 | <b>X</b><br>6-10am | <b>X</b><br>6-10am | | |
| NAbs | | | | <b>X</b><br>D30±5D | |
| Mortality (reason/diagnosis of death) | | | | x | x |
| Concomitant Medications/Therapies | • | ←X | | | |
| AE Recording | • | ←X> | | | |
| Deaths Recording | | x | | | |
| mRS | | | | | x |

#### KEY:

- \* Assessments prior to D30 are only performed if patient is still hospitalised in the same hospital initially operated. If the patient is moved to a different hospital, assessments will not be done. If study treatment is terminated early by Investigator decision due to patient improvement, the study assessment schedule should be followed as normal.
- \*\* From D6 to D30 assessment of vital signs, patient status and physical examination are performed as scheduled if hospitalised. Biochemistry, hematology, MxA, CD73 and PIM are assessed on D9 and D13 if patient is hospitalized. D9 to D30 assessments should be performed at the same time of day as D6 assessments. Note: Where a patient's condition precludes an assessment taking place as scheduled, the assessment should be performed within ± 2 hours of the scheduled time and if this is not possible, the assessment will not be performed and the reason for non-performance will be recorded.
- SOFA scores are assessed daily in the ICU from D0 pre-dose to D30, as applicable by standard clinical treatment at that point (therefore if a patient doesn't have an arterial line, no arterial blood sampling should be taken).

## Flow Chart for Discharge Prior to D30 and After D30

| 40050045450 | Withd | rawal |
|---|---|---|
| ASSESSMENTS | Prior to D30 | After D30 |
| Check whether the patient is in the ICU ❖ | X | X |
| Check whether the patient is on ventilation * | X | X |
| Check whether the patient is on organ support | X | X |
| SOFAs (the worst daily value should be used) | X | |
| Ventilator Free Days (VFDs) | X | |
| Physical Examination | X | |
| Vital Signs (Temp, BP, HR) | X | |
| Blood Biochemistry | X | |
| Haematology | X | |
| MxA, CD73 and PIM | х | |
| Days on Vasoactive Drugs | х | |
| Mortality (state the reason of death if possible)** | X | X |
| Concomitant Medications/Therapies | Х | |
| AE recording | х | |
| Death recording | Х | Х |

### KEY:

- ❖ Patients still on ICU who are transferred to another hospital or healthcare ICU facility prior to D30 are followed up to assess the days on ICU at scheduled D30 if applicable.
- \* Patients still on positive pressure ventilation who are transferred to another hospital or healthcare facility prior to D30 are followed up to assess the VFD outcome at scheduled D30.
- \*\* Mortality follow-up: For all patients, mortality is assessed at D90 (3 months). If a patient is lost to follow-up, when possible, mortality data will be sought from alternate sources such as the patient's local Physician or available national databases.

### Schedules for SOFAs

| | Baseline Period |
|-------------|-----------------|
| ASSESSMENTS | D0 pre-dose |
| SOFA | |

| | | | Treatmer | nt Period | | |
|-------------|--------------|----|----------|-----------|----|------------|
| ASSESSMENTS | D0 post dose | D1 | D2 | D3 | D4 | <b>D</b> 5 |
| SOFA | x | x | x | x | x | x |

| | | | | | | | | | | Ŋ, | Shor | t Te | rm F | ollo | w-Up | ) | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| ASSESSMENTS | D6 | D7 | D8 | D9 | D10 | D11 | D12 | D13 | D14 | D15 | D16 | D17 | D18 | D19 | D20 | D21 | D22 | D23 | D24 | D25 | D26 | D27 | D28. | D29 | D30 |
| SOFA | X | X | X | X | x | x | X | X | x | x | x | x | X | X | X | x | X | x | X | X | x | x | x | X | x |

# 19.3 Table and figure plan

| Demographic<br>Tables | |
|---|---|
| Table 14.1.1 | Disposition of patients |
| Table 14.1.2.1 | Demographics (categorical) (FAS-E) |
| Table 14.1.2.2 | Demographics (categorical) (PPS) |
| Table 14.1.3.1 | Demographics (continuous) (FAS-E) |
| Table 14.1.3.2 | Demographics (continuous) (PPS) |
| Table 14.1.4.1 | Major surgical outcomes affecting patient (FAS-E) |
| Table 14.1.4.2 | Major surgical outcomes affecting patient (PPS) |
| Table 14.1.5.1 | Surgical procedure and periprocedual information (FAS-E) |
| Table 14.1.5.2 | Surgical procedure and periprocedual information (FAS-E) |
| Table 14.1.6.1 | Medical history (FAS-E) |
| Table 14.1.6.2 | Medical history (PPS) |
| Table 14.1.7.1 | Concomitant medications/therapies (FAS-E) |
| Table 14.1.7.2 | Concomitant medications/therapies (PPS) |
| Table 14.1.8 | Pregnancy test (FAS-S) |
| <b>Efficacy Tables</b> | Efficacy |
| Table 14.2.1.1.1 | All-cause mortality D30 (FAS-E) |
| Table 14.2.1.1.2 | All-cause mortality D30 (PPS) |
| Table 14.2.1.2.1 | Logistic regression of All-cause mortality D30 (FAS-E) |
| Table 14.2.1.2.2 | Logistic regression of All-cause mortality D30 (PPS) |
| Table 14.2.1.3.1 | All-cause mortality D90 (FAS-E) |
| Table 14.2.1.3.2 | All-cause mortality D90 (PPS) |
| Table 14.2.1.4.1 | Cox regression of All-cause mortality D90 (FAS-E) |
| Table 14.2.1.4.2 | Cox regression of All-cause mortality D90 (PPS) |
| Table 14.2.1.5.1 | Logistic regression of All-cause mortality D90 (FAS-E) |
| Table 14.2.1.5.2 | Logistic regression of All-cause mortality D90 (PPS) |
| Table 14.2.1.6.1 | Number of VFDs up to D30 (FAS-E) |
| Table 14.2.1.6.2 | Number of VFDs up to D30 (PPS) |
| Table 14.2.1.7.1 | Number of ICU free days up to D30 (FAS-E) |
| Table 14.2.1.7.2 | Number of ICU free days up to D30 (PPS) |
| Table 14.2.1.8.1 | Organ failure free days up to D30 (FAS-E) |
| Table 14.2.1.8.2 | Organ failure free days up to D30 (PPS) |
| Table 14.2.1.9.1 | Number of days on hemodialysis up to D30 (FAS-E) |
| Table 14.2.1.9.2 | Number of days on hemodialysis up to D30 (PPS) |
| Table 14.2.1.9.3 | Number of days on hemodialysis up to D30 excluding deaths (FAS-E) |
| Table 14.2.1.9.4 | Number of days on hemodialysis up to D30 excluding deaths (PPS) |
| Table 14.2.1.10.1 | Number of days in hospital up to D30 (FAS-E) |
| Table 14.2.1.10.2 | Number of days in hospital up to D30 (PPS) |
| Table 14.2.1.10.3 | Number of days in hospital up to D30 excluding deaths (FAS-E) |
| Table 14.2.1.10.4 | Number of days in hospital up to D30 excluding deaths (PPS) |
| Table 14.2.1.11.1 | Length of stay in another health care facility up to D30 (FAS-E) |

| Table 14.2.1.11.2 | Length of stay in another health care facility up to D30 (PPS) |
|---|---|
| Table 14.2.1.11.3 | Length of stay in another health care facility up to D30 excluding deaths (FAS-E) |
| Table 14.2.1.11.4 | Length of stay in another health care facility up to D30 excluding deaths (PPS) |
| Table 14.2.1.12.1 | IAP values by timepoint (FAS-E) |
| Table 14.2.1.12.2 | IAP values by timepoint (PPS) |
| Table 14.2.1.12.3 | IAP values by timepoint excluding early deaths (FAS-E) |
| Table 14.2.1.12.4 | IAP values by timepoint excluding early deaths (PPS) |
| Table 14.2.1.13.1 | IAP grades by timepoint (FAS-E) |
| Table 14.2.1.13.2 | IAP grades by timepoint (PPS) |
| Table 14.2.1.13.3 | IAP grades by timepoint excluding early deaths (FAS-E) |
| Table 14.2.1.13.4 | IAP grades by timepoint excluding early deaths (PPS) |
| Table 14.2.1.14.1 | Disability on D90 measured with mRS (FAS-E) |
| Table 14.2.1.14.2 | Disability on D90 measured with mRS (PPS) |
| Table 14.2.1.14.1 | Neutralizing antibodies (FAS-E) |
| Table 14.2.1.14.2 | Neutralizing antibodies (PPS) |
| | Pharmacodynamics |
| Table 14.2.2.1.1 | MxA concentration (FAS-E) |
| Table 14.2.2.1.2 | MxA concentration (PPS) |
| Table 14.2.2.2.1 | MxA ANOVA (FAS-E) |
| Table 14.2.2.2.2 | MxA ANOVA (PPS) |
| Table 14.2.2.3.1 | CD73 concentration (FAS-E) |
| Table 14.2.2.3.2 | CD73 concentration (PPS) |
| Table 14.2.2.4.1 | CD73 ANOVA (FAS-E) |
| Table 14.2.2.4.2 | CD73 ANOVA (PPS) |
| Table 14.2.2.5.1 | Potential inflammatory markers (FAS-E) |
| Table 14.2.2.5.2 | Potential inflammatory markers (PPS) |
| Table 14.2.2.6.1 | PIM ANOVA (FAS-E) |
| Table 14.2.2.6.2 | PIM ANOVA (PPS) |
| | Subgroup analyses |
| Table 14.2.1.1.1 | All-cause mortality D30 by subgroups |
| Table 14.2.1.2.1 | Logistic regression of All-cause mortality D30 by subgroups |
| Safety Tables | |
| Table 14.3.1 | Extent of exposure and compliance (FAS-S) |
| Table 14.3.2 | Summary of TEAEs (FAS-S) |
| Table 14.3.3.1 | Treatment emergent adverse events (FAS-S) |
| Table 14.3.3.2 | TEAEs by causality (FAS-S) |
| Table 14.3.3.3 | TEAEs by severity (FAS-S) |
| Table 14.3.3.4 | TEAEs by maximum severity (FAS-S) |
| Table 14.3.3.5 | TEAEs by causality and severity (FAS-S) |
| Table 14.3.3.6 | TEAEs by causality and maximum severity (FAS-S) |
| Table 14.3.4.1 | TEAEs during treatment period (FAS-S) |
| Table 14.3.4.2 | TEAEs during treatment period by causality (FAS-S) |
| Table 14.3.4.3 | TEAEs during treatment period by severity (FAS-S) |

| Table 14.3.4.4 | TEAEs during treatment period by maximum severity (FAS-S) |
|---|---|
| Table 14.3.4.5 | TEAEs during treatment period by causality and severity (FAS-S) |
| Table 14.3.4.6 | TEAEs during treatment period by causality and maximum severity (FAS-S) |
| Table 14.3.5.1 | TEAEs during short-term follow-up period (FAS-S) |
| Table 14.3.5.2 | TEAEs during short-term follow-up period by causality (FAS-S) |
| Table 14.3.5.3 | TEAEs during short-term follow-up period by severity (FAS-S) |
| Table 14.3.5.4 | TEAEs during short-term follow-up period by maximum severity (FAS-S) |
| Table 14.3.5.5 | TEAEs during short-term follow-up period by causality and severity (FAS-S) |
| Table 14.3.5.6 | TEAEs during short-term follow-up period by causality and maximum severity (FAS- |
| 14010 14.3.3.0 | S) |
| Table 14.3.6 | Listing of other adverse events (FAS-S) |
| Table 14.3.7 | TEAEs leading to discontinuation (FAS-S) |
| Table 14.3.8 | Serious TEAES (FAS-S) |
| Table 14.3.9.1 | Biochemistry - Descriptive statistics (FAS-S) |
| Table 14.3.9.2 | Biochemistry - Categorical analysis (FAS-S) |
| Table 14.3.9.3 | Biochemistry - Shift tables (FAS-S) |
| Table 14.3.10.1 | Haematology - Descriptive statistics (FAS-S) |
| Table 14.3.10.2 | Haematology - Categorical analysis (FAS-S) |
| Table 14.3.10.3 | Haematology - Shift tables (FAS-S) |
| Table 14.3.11.1 | Vital signs - Descriptive statistics (FAS-S) |
| Table 14.3.11.2 | Vital signs - Change from baseline (FAS-S) |
| Table 14.3.11.3 | Vital signs - Maximum change from baseline (FAS-S) |
| Table 14.3.12.1 | Physical examination (FAS-S) |
| Table 14.3.12.2 | Physical examination - Shift from screening to D30 |

# 19.4 Data listing plan

| Listing 16.2.1 | Disposition of subjects |
|-----------------|-----------------------------------------------------------|
| Listing 16.2.2 | Study discontinuations |
| Listing 16.2.3 | Extent of exposure |
| Listing 16.2.4 | Drug accountability |
| Listing 16.2.5 | Inclusion/exclusion criteria |
| Listing 16.2.6 | Demographic and other baseline characteristics |
| Listing 16.2.7 | Medical history and concomitant diseases |
| Listing 16.2.8 | Prior and concomitant medications/therapies |
| Listing 16.2.9 | Major surgical outcomes affecting patient |
| Listing 16.2.10 | Surgical procedure and peri procedual information |
| Listing 16.2.11 | Pregnancy test results |
| Listing 16.2.12 | Clinical event data |
| Listing 16.2.13 | Death and reasons for death |
| Listing 16.2.14 | Daily status data |
| Listing 16.2.15 | All-cause mortality data |
| Listing 16.2.16 | Number of VFD and ICU free days |
| Listing 16.2.17 | Length of stay in hospital and other health care facility |
| Listing 16.2.18 | Number of days in hemodialysis |
| Listing 16.2.19 | MxA and CD73 concentration data |
| Listing 16.2.20 | Potential inflammatory markers data |
| Listing 16.2.21 | Neutralizing antibodies data |
| Listing 16.2.22 | Intra-abdominal pressure data |
| Listing 16.2.23 | Disability measured with mRS |
| Listing 16.2.24 | SOFA score data |
| Listing 16.2.25 | Non-treatment emergent adverse events |
| Listing 16.2.26 | Treatment emergent adverse events |
| Listing 16.2.27 | Serious adverse events |
| Listing 16.2.28 | Adverse events leading to discontinuation |
| Listing 16.2.29 | Biochemistry data |
| Listing 16.2.30 | Haematology data |
| Listing 16.2.31 | Vital signs data |
| Listing 16.2.32 | Physical examination data |